CLINICAL TRIAL: NCT01124110
Title: Tobacco Tactics Website for Operating Engineers
Acronym: BCBSM-OE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Sonia Duffy, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N011646 - 1465.RFP
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Smoking; Tobacco Use Cessation
Keywords: Operating Engineers; Smoking Cessation
MeSH Terms: conditions — Smoking; Tobacco Use Cessation; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1-800-QUIT-NOW Telephone Hotline (Other): The control group receives efficacious smoking cessation treatment via the 1-800-QUIT-NOW telephone hotline. The 1-800-QUIT-NOW hotline is a national program. The first time smokers call the hotline, they receive a personal coach who assists them in setting a quit date and making an individualized quit plan. The personal coach also provides on-going support with up to five telephone coaching sessions around the caller's quit date.
  Interventions: Other: 1-800-QUIT-NOW Telephone Hotline
- Tobacco Tactics Intervention (Experimental): This intervention contains a website, medications, and nurse counseling.
  Interventions: Behavioral: Tobacco Tactics Web-Based Intervention

INTERVENTIONS:
Behavioral: Tobacco Tactics Web-Based Intervention — The Tobacco Tactics Web-Based Intervention contains website, medications, and nurse counseling.
  Arms: Tobacco Tactics Intervention
Other: 1-800-QUIT-NOW Telephone Hotline — The control group receives efficacious smoking cessation treatment via the 1-800-QUIT-NOW telephone hotline. The 1-800-QUIT-NOW hotline is a national program. The first time smokers call the hotline, they receive a personal coach who assists them in setting a quit date and making an individualized quit plan. The personal coach also provides on-going support with up to five telephone coaching sessions around the caller's quit date.
  Arms: 1-800-QUIT-NOW Telephone Hotline

SUMMARY:
This is a clustered randomized control trial to test the Tobacco Tactics intervention among Operating Engineers (heavy equipment workers). The intervention group will be directed to the Tobacco Tactics website, and the control group will be directed to the state supported 1-800 quit-now telephone hotline during routine annual safety training that all Operating Engineers are required to attend. The web-based quitting intervention includes provision of over-the-counter nicotine replacement therapy and will be followed by nurse email and/or telephone counseling. It is expected that Operating Engineers who are randomized to the Tobacco Tactics website intervention will have at least equal or greater decreases in smoking at 30-day and 6-month follow-up compared to those randomized to the 1-800-QUIT-NOW quit line. In addition, the investigators expect to find that Operating Engineers randomized to the Tobacco Tactics website intervention will: a) be able to accomplish tasks; b) be able to accomplish goals with skill and speed; c) be able to operate the system; d) be satisfied with the website; e) access the site repeatedly; and f) spend time on the site during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* attending a training session provided by the Operating Engineers Local 324 Education Center
* greater than 18 years of age
* smoked cigarettes in the past month
* interested in participating in a program to quit smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2010-01; Primary Completion 2013-03 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Quit Rate | 30-day Follow-Up
  The investigators will measure 7-day point prevalence abstinence by asking the well validated question, "Have you used any tobacco products (even one puff) in the past 7 days?" The investigators will also assess harm reduction (ability to quit at all, number of quit attempts, and number of cigarettes smoked per day).
Quit Rate | 6-Month Follow-Up
  The investigators will measure 7-day point prevalence abstinence by asking the well validated question, "Have you used any tobacco products (even one puff) in the past 7 days?" Smoking status will be confirmed by biochemical verification in the form of urinary cotinine test strips. The investigators will also assess harm reduction (ability to quit at all, number of quit attempts, and number of cigarettes smoked per day).

CONTACTS AND LOCATIONS:
Overall Officials: Sonia A Duffy, PhD, RN, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, School of Nursing, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Fiore MC. US public health service clinical practice guideline: treating tobacco use and dependence. Respir Care. 2000 Oct;45(10):1200-62. PMID 11054899
- [Background] Solomon LJ, Scharoun GM, Flynn BS, Secker-Walker RH, Sepinwall D. Free nicotine patches plus proactive telephone peer support to help low-income women stop smoking. Prev Med. 2000 Jul;31(1):68-74. doi: 10.1006/pmed.2000.0683. PMID 10896845
- [Background] Rice VH, Stead LF. Nursing interventions for smoking cessation. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD001188. doi: 10.1002/14651858.CD001188.pub3. PMID 18253987
- [Background] Lichtenstein E, Glasgow RE, Lando HA, Ossip-Klein DJ, Boles SM. Telephone counseling for smoking cessation: rationales and meta-analytic review of evidence. Health Educ Res. 1996 Jun;11(2):243-57. doi: 10.1093/her/11.2.243. PMID 10163409
- [Background] Stern F, Haring-Sweeney M. Proportionate mortality among unionized construction operating engineers. Am J Ind Med. 1997 Jul;32(1):51-65. doi: 10.1002/(sici)1097-0274(199707)32:13.0.co;2-u. PMID 9131212
- [Background] Lee DJ, Fleming LE, McCollister KE, Caban AJ, Arheart KL, LeBlanc WG, Chung-Bridges K, Christ SL, Dietz N, Clark JD 3rd. Healthcare provider smoking cessation advice among US worker groups. Tob Control. 2007 Oct;16(5):325-8. doi: 10.1136/tc.2006.019117. PMID 17897991
- [Background] Moher M, Hey K, Lancaster T. Workplace interventions for smoking cessation. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD003440. doi: 10.1002/14651858.CD003440.pub2. PMID 15846667
- [Background] Lenert L, Munoz RF, Stoddard J, Delucchi K, Bansod A, Skoczen S, Perez-Stable EJ. Design and pilot evaluation of an internet smoking cessation program. J Am Med Inform Assoc. 2003 Jan-Feb;10(1):16-20. doi: 10.1197/jamia.m1128. PMID 12509354
- [Derived] Choi SH, Waltje AH, Ronis DL, Noonan D, Hong O, Richardson CR, Meeker JD, Duffy SA. Web-enhanced tobacco tactics with telephone support versus 1-800-QUIT-NOW telephone line intervention for operating engineers: randomized controlled trial. J Med Internet Res. 2014 Nov 20;16(11):e255. doi: 10.2196/jmir.3375. PMID 25447467
- [Derived] Duffy SA, Ronis DL, Richardson C, Waltje AH, Ewing LA, Noonan D, Hong O, Meeker JD. Protocol of a randomized controlled trial of the Tobacco Tactics website for operating engineers. BMC Public Health. 2012 May 17;12:335. doi: 10.1186/1471-2458-12-335. PMID 22569211
- See also: Front Page of the Tobacco Tactics Website — http://bcbsm-operatingengineers.nursing.umich.edu/